CLINICAL TRIAL: NCT01114412
Title: Description of Basic Visceral Sensations Coming From the Bladder
Brief Title: Basic Sensations Coming From the Bladder
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-4-045.8
Record Dates: First submitted 2010-04-29; First posted 2010-05-03 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2010-04

CONDITIONS: Healthy; Overactive Bladder Syndrome
Keywords: focus groups; overactive bladder; bladder sensations
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with overactive bladder syndrome
- Healthy volunteers: Healthy volunteers

SUMMARY:
A major complication in studies to identify the nature of bladder sensations is language. It is difficult, if not near impossible, for the lay person, with no knowledge of physiology, anatomy or pathology, to put into simple terms a description of basic visceral sensations. Therefore, before the investigators can speculate about the detailed mechanisms generating sensation the investigators must overcome this language and communication difficulty. This will be addressed in the present study.

There are important reasons why the investigators must identify the mechanisms generating the different sensations as the bladder fills. One of them is that these are basic physiological mechanisms which need to be better understood.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers

* Healthy students from The University of Maastricht well versed in Dutch.

Patients

* Patients with OAB diagnosed by their urologist using the criteria of more than 8 micturitions on three consecutive days. Before the start of any anticholinergic or other therapy. Patients on anticholinergic therapy will be asked to stop this therapy for at least 10 days before they enter the first session.
* Well versed in Dutch.

Exclusion Criteria:

Healthy volunteers

* Use of any medication (except oral contraceptives)
* Surgical history of the abdomen
* Urinary complaints (e.g. frequency, urgency)
* Urinary tract infection

Patients:

* Congestive heart disease or history of heart failure
* Presence of urinary tract infection. These patients will be treated by antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
  Patients with overactive bladder
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
description of bladder sensations
  The primary objective of this experiment is to address how medical students and patients with OAB describe the sensations they feel during the filling phase of the bladder.
  Primary objectives
  * To put into simple terms a description of basic visceral sensations coming from the bladder
  * Describe the pattern of normal sensations during filling

CONTACTS AND LOCATIONS:
Overall Officials: Gommert A van Koeveringe, MD, PhD, Urologist, Study Director — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands